CLINICAL TRIAL: NCT01648231
Title: An Open-label, Randomized, Single Dose, Three-way Crossover Study to Determine the Comparative Bioavailability of Two Fixed Dose Combination Tablet Formulations of Amlodipine (5mg) and Losartan (100mg) in Healthy Adult Male and Female Subjects Under Fasting Conditions
Brief Title: Crossover Study to Evaluate the Comparative Bioavailability of Two Fixed Dose Combination Tablet Formulations of Amlodipine and Losartan in Health Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 116797
Record Dates: First submitted 2012-07-12; First posted 2012-07-24 (Estimated); Last update posted 2017-07-26 (Actual); Status verified 2017-07

CONDITIONS: Hypertension
Keywords: Healthy Volunteer
MeSH Terms: conditions — Hypertension | interventions — Amlodipine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Treatment Period 1 (Other): 1 x 5mg amlodipine tablet and 1 x 100mg losartan tablet administered in fasted state
  Interventions: Drug: Reference Treatment: 1 x 5mg amlodipine tablet and 1 x 100mg losartan tablet administered in fasted state
- Treatment Period 2 (Other): 1 x 5mg amlodipine / 100mg losartan tablet administered in fasted state
  Interventions: Drug: Fixed Dose Combination 1: 1 x 5mg amlodipine / 100mg losartan tablet administered in fasted state
- Treatment Period 3 (Other): 1 x 5mg amlodipine / 100mg losartan tablet administered in fasted state
  Interventions: Drug: Fixed Dose Combination 2: 1 x 5mg amlodipine / 100mg losartan tablet administered in fasted state

INTERVENTIONS:
Drug: Reference Treatment: 1 x 5mg amlodipine tablet and 1 x 100mg losartan tablet administered in fasted state — 1 x 5mg amlodipine tablet and 1 x 100mg losartan tablet administered in fasted state
  Other Names: GSK2944406
  Arms: Treatment Period 1
Drug: Fixed Dose Combination 1: 1 x 5mg amlodipine / 100mg losartan tablet administered in fasted state — 1 x 5mg amlodipine / 100mg losartan tablet administered in fasted state
  Other Names: GSK2944406
  Arms: Treatment Period 2
Drug: Fixed Dose Combination 2: 1 x 5mg amlodipine / 100mg losartan tablet administered in fasted state — 1 x 5mg amlodipine / 100mg losartan tablet administered in fasted state
  Other Names: GSK2944406
  Arms: Treatment Period 3

SUMMARY:
The purpose of this study is to evaluate the comparative bioavailability of two fixed dose combination tablet formulations of amlodipine and losartan in healthy volunteers. Subjects will receive each of the following three treatments administered in a randomized three-way crossover design: a reference treatment consisting of a 5mg amlodipine tablet and 100mg losartan tablet; a fixed dose combination tablet consisting of 5mg amlodipine and 100mg losartan; and another fixed dose combination tablet consisting of 5mg amlodipine and 100mg losartan; all three treatments will be administered once orally and in a fasted state. Serial blood samples will be obtained at pre-defined timepoints for pharmacokinetic analysis of amlodipine, losartan and carboxylic acid (this is the primary active losartan metabolite). Safety assessments will include measurements of orthostatic vital signs, electrocardiograms (ECG), collection of adverse events (AE) and clinical laboratory tests.

DETAILED DESCRIPTION:
Amlodipine and losartan are calcium channel and angiotensin II receptor type-1 blockers, respectively, and are established treatments to manage blood pressure (BP) levels for patients with hypertension; both medications are currently marketed in the United States and Europe as anti-hypertensive agents. This is a an open-label, randomized, single dose, three-way crossover study enrolling 24 healthy adult male and female subjects under fasting conditions. Each subject will participate in three treatment periods. The study consists of a screening phase, three treatment periods and a follow-up visit. Subjects will receive each of the following three treatments administered in a randomized three-way crossover design: a reference treatment consisting of a single 5mg amlodipine tablet and a single 100mg losartan tablet; a single fixed dose combination tablet consisting of 5mg amlodipine and 100mg losartan; and another single fixed dose combination tablet consisting of 5mg amlodipine and 100mg losartan; all three treatments will be administered once orally and in a fasted state. Serial blood samples will be obtained at pre-defined timepoints for pharmacokinetic analysis of amlodipine, losartan and carboxylic acid (this is the primary active losartan metabolite). Safety assessments will include measurements of orthostatic vital signs, electrocardiograms (ECG), collection of adverse events (AE) and clinical laboratory tests.

ELIGIBILITY:
Inclusion Criteria:

* Male or female between 18 and 65 years of age inclusive, at the time of signing the informed consent.
* Alanine transaminase (ALT), alkaline phosphatase and bilirubin ≤ 1.5 x upper limit of normal (ULN; isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%)
* Normal electrocardiogram (ECG) morphology and measurements. In particular QTc <450 msec or QT < 480 msec in subjects with Bundle Branch Block based on an average from three ECGs obtained over a brief recording period.
* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring. A subject with a clinical abnormality or laboratory parameters outside the reference range for the population being studied may be included only if the Investigator feels that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures..
* A female subject is eligible to participate if she is of:

Non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea (in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) > 40 MlU/ml and estradiol < 40 pg/ml (<147 pmol/L) is confirmatory. Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use a protocol approved contraception method if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrollment. For mostforms of HRT, at least 2-4 weeks will elapse between the cessation of therapy and the blood draw; this interval depends on the type and dosage of HRT. Following confirmation of their post-menopausal status, they can resume use of HRT during the study without use of a contraceptive method.

Child-bearing potential and agrees to use one of the protocol approved contraception methods for an appropriate period of time (as determined by the product label or investigator) prior to the start of dosing to sufficiently minimize the risk of pregnancy at that point. Female subjects must agree to use contraception until 14 days post-last dose of amlodipine/losartan.

* Body weight ≥ 50 kg and a body mass index (BMI) within the range 19 - 32 kg/m2 (inclusive).
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.

Exclusion Criteria:

* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening.
* Any subject with a systolic blood pressure (BP) <95mmHg or with a recent history of postural symptoms.
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* A positive pre-study drug/alcohol screen.
* A positive test for HIV antibody.
* History of regular alcohol consumption within 6 months of the study defined as:

An average weekly intake of >21 units for males or >14 units for females. One unit is equivalent to 8 g of alcohol: a half-pint (~240 ml) of beer, 1 glass (100 ml) of wine or 1 (25 ml) measure of spirits.

* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day
* Unable to refrain from the use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* Pregnant females as determined by positive urine human chorionic gonadotrophin (hCG) test at Day -1 or serum hCG at all other timepoints.
* Lactating females.
* Unwillingness or inability to follow the procedures outlined in the protocol.
* Subject is mentally or legally incapacitated.
* History of sensitivity to heparin or heparin-induced thrombocytopenia.
* Subjects who have asthma or a history of asthma
* Urinary cotinine levels indicative of smoking or history or regular use of tobacco- or nicotine-containing products within 6 months prior to screening.
* Positive carbon monoxide (CO) on admission to the Unit.
* Unable to refrain from consumption of red wine, seville oranges, grapefruit or grapefruit juice (and/or pummelos, exotic citrus fruits, grapefruit hybrids or fruit juices) from 7 days prior to the first dose of study medication.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2012-08-06 (Actual); Primary Completion 2012-09-25 (Actual); Study Completion 2012-09-25 (Actual)

PRIMARY OUTCOMES:
Plasma concentration of amlodipine and losartan: Peak plasma concentration (Cmax) and last measurable plasma concentration (Clast) | Participants will be followed and monitored for the duration of their hospital stay (24 hours per treatment period). The longest duration of participation in the study will be approximately 14 weeks
  Comparison of Cmax and Clast after administration of two amlodipine and losartan fixed dose combinations in comparison to reference treatment (to determine the comparative bioavailability)
Time to peak plasma concentration (Tmax) of amlodipine and losartan | Participants will be followed and monitored for the duration of their hospital stay (24 hours per treatment period). The longest duration of participation in the study will be approximately 14 weeks
  Comparison of Tmax after administration of two amlodipine and losartan fixed dose combinations in comparison to reference treatment (to determine the comparative bioavailability)
Area under the plasma concentration-time curve (AUC) of amlodipine and losartan: from time zero to time t (AUCt), from time zero to infinity (AUCinf) and time t to infinity as a percentage of total AUC (%AUCex) | Participants will be followed and monitored for the duration of their hospital stay (24 hours per treatment period). The longest duration of participation in the study will be approximately 14 weeks
  Comparison of AUCt, AUCinf and %AUCex after administration of two amlodipine and losartan fixed dose combinations in comparison to reference treatment (to determine the comparative bioavailability)
Elimination half-life (t½) of amlodipine and losartan | Participants will be followed and monitored for the duration of their hospital stay (24 hours per treatment period). The longest duration of participation in the study will be approximately 14 weeks
  Comparison of t½ after administration of two amlodipine and losartan fixed dose combinations in comparison to reference treatment (to determine the comparative bioavailability)

SECONDARY OUTCOMES:
Number of healthy volunteers with adverse events | Participants will be followed and monitored for the duration of their hospital stay (24 hours per treatment period). The longest duration of participation in the study will be approximately 14 weeks
  Comparison of adverse events (as determined by orthostatic vital sign and electrocardiogram measurements and clinical lab results) after administration of two amlodipine and losartan fixed dose combinations in comparison to reference treatment (to determine the safety and tolerability)
Plasma concentration of of carboxylic acid: Peak plasma concentration (Cmax) | Participants will be followed and monitored for the duration of their hospital stay (24 hours per treatment period). The longest duration of participation in the study will be approximately 14 weeks
  Comparison of Cmax and Clast after administration of two amlodipine and losartan fixed dose combinations in comparison to reference treatment (to determine the comparative bioavailability)
Elimination half-life (t½) of carboxylic acid | Participants will be followed and monitored for the duration of their hospital stay (24 hours per treatment period). The longest duration of participation in the study will be approximately 14 weeks
  Comparison of t½ after administration of two amlodipine and losartan fixed dose combinations in comparison to reference treatment (to determine the comparative bioavailability)
Time to peak plasma concentration (Tmax) of carboxylic acid | Participants will be followed and monitored for the duration of their hospital stay (24 hours per treatment period). The longest duration of participation in the study will be approximately 14 weeks
  Comparison of Tmax after administration of two amlodipine and losartan fixed dose combinations in comparison to reference treatment (to determine the comparative bioavailability)
Area under the plasma concentration-time curve (AUC) of carboxylic acid: from time zero to time t (AUCt), from time zero to infinity (AUCinf) and time t to infinity as a percentage of total AUC (%AUCex) | Participants will be followed and monitored for the duration of their hospital stay (24 hours per treatment period). The longest duration of participation in the study will be approximately 14 weeks
  Comparison of AUCt, AUCinf and %AUCex after administration of two amlodipine and losartan fixed dose combinations in comparison to reference treatment (to determine the comparative bioavailability)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Randwick, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- See also: Results for study 116797 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/116797?search=study&search_terms=116797#rs
- Available data/document: Statistical Analysis Plan: 116797 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 116797 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 116797 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 116797 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 116797 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 116797 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 116797 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register